CLINICAL TRIAL: NCT06664528
Title: Cardiovascular Health and Prognosis in Adult Patients With Cancer Exposed to Cardiotoxic Therapies, an Observational Study
Brief Title: Cardiovascular Health in Adult Patients With Cancer Exposed to Cardiotoxic Therapies
Acronym: CV_CANCER
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6977
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Toxicity; Cancer
MeSH Terms: conditions — Cardiotoxicity; Neoplasms | interventions — Echocardiography; Electrocardiography; Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECHOCARDIOGRAPHY — A complete echocardiographic exam will be performed during each cardio-oncologic evaluation.
Diagnostic Test: ELECTROCARDIOGRAPHY (ECG) — An ECG tracing will be obtained during each cardio-oncologic evaluation.
Diagnostic Test: LABORATORY TESTS — The cardiac biomarkers high-sensitivity troponin I and N-terminal pro-B-type natriuretic peptide (NT-proBNP) will be dosed according to the current recommendations of Cardio-Oncology Guidelines.

SUMMARY:
The goal of this observational study is to evaluate the cardiovascular health and prognosis of adult patients with cancer, treated with cardiotoxic therapies.

The main purposes of the study are the following:

* Identify the demographic factors related to the onset of cardiotoxicity produced by anticancer drugs.
* Identify any subgroups more likely to develop distant major adverse cardiovascular events (MACE).
* Evaluate the usefulness of clinical, biohumoral and echocardiographic parameters for early diagnosis of cardiotoxicity.

Participants will be monitored during the anticancer treatment via clinical, laboratory and instrumental evaluation according to the recommendation of the current guidelines on Cardio-Oncology (European Society of Cardiology, 2022). Initial follow-up will be 2 years.

DETAILED DESCRIPTION:
The goal of this observational study is to evaluate the cardiovascular health and prognosis of adult patients with cancer, exposed to potentially-cardiotoxic therapies.

The main purposes of the study are the following:

* Identify the demographic factors related to the onset of cardiotoxicity produced by anticancer drugs.
* Identify any subgroups of patients more likely to develop distant major adverse cardiovascular events (MACE).
* Evaluate the usefulness of clinical, bio-humoral and echocardiographic parameters for early diagnosis of cardiotoxicity.

Participants will be monitored during the anticancer treatment via clinical, laboratory and instrumental evaluation according to the recommendations of the available guidelines on Cardio-Oncology (European Society of Cardiology, 2022). Initial follow-up will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 at the time of evaluation
* Patients treated with potentially cardiotoxic anticancer drugs
* Patients for which complete clinical, electrocardiographic and echocardiographic data are available at first evaluation and at least at one follow-up visit.

Exclusion Criteria:

* Patients under the age of 18 at the time of evaluation
* Patients whose documentation of the first visit is not available
* Patients for whom it is not possible to obtain follow-up information through a medical visit or by telephone
* Patient with poor acoustic window for echocardiographic examination.
* Refusal of informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cancer treated with potentially cardiotoxic anticancer drugs, with complete clinical, laboratory, electrocardiographic and echocardiographic data obtained at the first cardio-oncologic evaluation and at least at one follow-up visit.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiotoxicity | 24 months
  Incidence of cancer therapy-related cardiovascular toxicity according to the definitions of the European Society of Cardiology Cardio-Oncology Guidelines, published in 2022.
Identification of major cardiovascular adverse events (MACE) | 24 months
  Identification of cardiovascular death, non-cardiovascular death and hospitalization for cardiac causes (congestive heart failure, major arrhythmias) both during the antineoplastic treatments and in the long-survivors population.

SECONDARY OUTCOMES:
Identification of early predictors of cardiotoxicity | 24 months
  Identification of any anamnestic, clinical, electrocardiographic and echocardiographic predictors of cardiotoxicity or major cardiovascular adverse events (MACE) at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Lombardo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS;UOSD diagnostica cardiologica non invasiva, Rome, Lazio, Italy